CLINICAL TRIAL: NCT00044434
Title: Bupropion as a Smoking Cessation Aid in Alcoholics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAGRA13689
Record Dates: First submitted 2002-08-28; First posted 2002-08-30 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Alcoholism; Smoking
MeSH Terms: conditions — Alcoholism; Smoking | interventions — Bupropion

INTERVENTIONS:
Drug: bupropion (Wellbutrin)

SUMMARY:
The purpose of this study is to test the use of time-released bupropion (Wellbutrin) in patients receiving treatment for alcohol abuse/dependence as an aid to stop smoking. Patients will receive either a time-released bupropion or placebo. Both groups will receive nicotine replacement therapy during the 9 week study. A final followup assessment will be conducted 6 months from the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Currently a patient in the Omaha VA Medical Center, Substance Abuse Treatment Center (SATC) or at Catholic Charities Campus for Hope.
* Have a diagnosis of alcohol abuse or alcohol dependence.
* Smoke 20 or more cigarettes/day (may also smoke pipes/cigars).
* Be interested in quitting smoking.
* Provide name, addresses, and phone numbers of at least two individuals who can provide information on their alcohol, nicotine, and other drug use during the follow-up period.
* If female, patient must a) be of non-childbearing potential, b) have a negative pregnancy test, c) sign a document stating they do not plan on becoming pregnant during the study.
* Agree to sign informed consent.
* Able to read and understand study-related forms and procedures.

Exclusion Criteria:

* Advanced cardiac, pulmonary, renal, or liver disease.
* History of seizures.
* History of brain tumor or significant head trauma.
* History of bulimia or anorexia nervosa.
* Current major depressive disorder or past history of panic disorders, schizophrenia, or bipolar affective disorder.
* Using psychoactive drugs.
* Receiving treatment with medications that lower seizure thresholds.
* Use of an investigational drug in any study in the past four weeks.
* Currently using any asthma medication.
* Used time-released bupropion in the past 12 months.
* Currently using any other treatments to stop smoking.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-05; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA/Nebraska/Western Iowa Health Care System, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961